CLINICAL TRIAL: NCT04213677
Title: Efficacy and Safety of Dapagliflozin in Polycystic Ovary Syndrome: a Multicentre, Randomized, Placebo-controlled Trial
Brief Title: Dapagliflozin Efficacy and Action in PCOS
Acronym: DEAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Huijie Zhang, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFEC-2019-243
Record Dates: First submitted 2019-12-04; First posted 2019-12-30 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; SGLT2 inhibitor
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin (Participants will receive dapagliflozin 10mg po qd).
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo (Participants will receive placebo po qd)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Participants will receive dapagliflozin 10mg po qd. Additionally, participants will receive lifestyle modification and nutrition education.
  Arms: Dapagliflozin
Drug: Placebo — Participants will receive placebo po qd. Additionally, participants will receive lifestyle modification and nutrition education.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of dapagliflozin on improving insulin resistance and hyperandrogenemia in obesity women with polycystic ovary syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. women aged 18 to 45 years;
2. Subjects with PCOS diagnosed by according to the Rotterdam criteria;
3. BMI ≥24 kg/m2 and/ or Homeostatic model assessment of insulin resistance (HOMA-IR) with a cutoff ≥2.5;
4. No pregnancy plan within the next 6 months;

Exclusion Criteria:

1. Congenital adrenal hyperplasia such as 21-hydroxylase deficiency, hyperprolactinemia, Cushing syndrome, androgen-producing tumors of the adrenal gland or ovary;
2. Other endocrine diseases include poorly controlled thyroid diseases (hyperthyroidism or hypothyroidism), acromegaly, type 2 diabetes;
3. Patients with a history of acute / chronic infection, severe cardio-cerebrovascular diseases and acute / chronic pancreatitis;
4. Taking any antidiabetic medication that would affect insulin resistance or hyperandrogenemia (i.e. TZD, GLP-1RA, DPP-4i, metformin) in the past one month;
5. Taking letrozole, clomiphene, oral contraceptive, glucocorticoid, gonadotropin, gonadotropin releasing hormone agonist, anti-androgen drug (spironolactone, cycloproterenone acetate, Flutamide etc.) and/or other drugs for PCOS in the past three months;
6. History of recurrent urinary tract infection;
7. History of malignant tumor;
8. Currently participating in weight loss programs or weight change in the past 3 months (> 5% current body weight) or have a history of gastrointestinal surgery.
9. Serious liver dysfunction or chronic kidney disease (AST or ALT > 3 times the upper limit of normal, or eGFR<30 ml/min/1.73 m2);
10. Women who are pregnant or plan to become pregnant;
11. Subject is, in the judgment of the Investigator, unlikely to comply with the protocol or has any severe concurrent medical or psychological condition that may affect the interpretation of efficacy or safety data;
12. Participation in other clinical trial in the 4 weeks before randomization;
13. Patients who are unwilling or unable to give informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Improvement in insulin resistance over 12 weeks | Baseline and 12 weeks
  Change in insulin resistance assessed by insulin sensitivity index(HOMA-IR)
Improvement in serum androgen level over 12 weeks | Baseline and 12 weeks
  Change in androgen level assessed by free testosterone index(FAI)

SECONDARY OUTCOMES:
Change in AUC (area under a curve) of glucose and insulin during the oral glucose tolerant test (OGTT) | Baseline to 12 week
Change in serum free testosterone(FT) | Baseline to 12 week
Change in serum sex hormone binding globulin(SHBG) | Baseline to 12 week
Net change in total testosterone (TT) level | Baseline and 12 weeks
Net change in dehydroepiandrosterone-sulfate(DHEAS) level | Baseline and 12 weeks
Net change in androstenedione(AD) level | Baseline and 12 weeks
Net change in luteinzing hormone(LH) level | Baseline and 12 weeks
Net change in waist circumference | Baseline to 12 week
Net Change in liver fat | Baseline to 12 week
  Liver fat will be assessed by liver fibroscan.
Change in ovulation rate assessed by serum progesterone | Baseline to 12 week
Net change in body weight | Baseline to 12 week
Net change in BMI | Baseline to 12 week
Net change in glucose | Baseline to 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China